CLINICAL TRIAL: NCT05526170
Title: Personalized Detection of Triggers and Risk Factors for Recurrence of Atrial Fibrillation and Other Atrial Arrhythmias With the Use of Long-term Monitoring
Brief Title: Triggers and Risk Factors for Recurrence of Atrial Arrhythmias With the Use of Long-term Monitoring
Acronym: TriggersAF
Status: Active, not recruiting | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: TriggersAF
Record Dates: First submitted 2022-02-17; First posted 2022-09-02 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Atrial Arrhythmia; Atrial Tachycardia; Premature Atrial Contractions; Arterial Hypertension; Sleep Disorder; Sleep Apnea; Stress; Physical Inactivity; Overexertion; Alcohol Drinking; Caffeine Dependence
Keywords: Atrial Fibrillation; Atrial Flutter; Atrial Arrhythmias; Arterial Hypertension; Triggers; Sleep disorders; Sleep apnea; Telemedicine; Mhealth; Remote monitoring; Digital health
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Atrial Premature Complexes; Hypertension; Sleep Wake Disorders; Sleep Apnea Syndromes; Sedentary Behavior; Alcohol Drinking | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with previously diagnosed paroxysmal or persistent atrial fibrillation: Patients with previously diagnosed paroxysmal or persistent atrial fibrillation who are in sinus rhythm at inclusion time. During trial period subjects will be monitored for different atrial arrhythmias and divided into the following subgroups: atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions (bigeminy, trigeminy, couplets), multiple atrial arrhythmias and no arrhythmia detected.
  Interventions: Device: Devices for long-term monitoring of objective and subjective parameters of the body

INTERVENTIONS:
Device: Devices for long-term monitoring of objective and subjective parameters of the body — Patients will use a 1-lead Holter ECG (Bittium Faros) for heart rhythm and physical activity analysis, a wearable wrist-worn device with photoplethysmography and 6-lead ECG for heart rhythm analysis, a sleep tracking mat (Withings sleep analyser) for sleep analysis, a smartphone with triggers application for entering the subjective triggers (stress, coffee, alcohol intake and others), a 48-hour ambulatory blood pressure monitor for 2 days and a regular blood pressure monitor for up to 5 days. Patients will be monitored for up to 7 days with the described system of devices. In addition, patients will receive investigations of heart echocardiography, laboratory tests and surveys to evaluate the system and the use of acquired information.

SUMMARY:
A prospective cohort study to evaluate the association between various triggers encountered in daily life and induction of atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia and premature atrial contractions) with the use of long-term monitoring devices. The collected data of personalized triggers and risk factors will be used to define the individual phenotype of atrial arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously diagnosed paroxysmal or persistent atrial fibrillation who are in sinus rhythm at inclusion time.
* An informed consent is signed by the patient.

Exclusion Criteria:

* The qualifying episode of AF has never been documented in ECG or Holter ECG monitoring.
* Patients with atrial fibrillation, atrial flutter or atrial tachycardia at inclusion time.
* Patients with permanent atrial fibrillation or permanent atrial flutter.
* Age <18 years.
* Patients with a pacemaker or an implanted cardiovert-defibrillator.
* Patients suffering from dementia or other severe neurological disorders and thus incapable to participate.
* Patients who present with antisocial behavior and/or do not want to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously diagnosed paroxysmal or persistent atrial fibrillation who are in sinus rhythm at inclusion time.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure association with atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 7 days
  Patterns of blood pressure fluctuations in relation to atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a monitoring period of 7 days. An association between episodes of uncontrolled arterial hypertension and occurrence of arrhythmia episodes is anticipated.

SECONDARY OUTCOMES:
Association of various triggers with atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 7 days
  Patterns of distinct triggers in relation to atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a monitoring period of 7 days. Mobile application and accelerometer of Holter ECG device will be used to record these factors as well as mark the time and the frequency of these actions. Attempts will be made to link all patient-marked triggers, their frequency, time of onset to the occurrence of arrhythmia.
  Triggers such as:
  coffee intake alcohol consumption distinguished by strength into:
  * spirits: brandy, vodka,
  * vine or champagne
  * low alcohol drinks: beer, cider emotional stress, overeating, physical activity, strenuous exercise, cold food, cold drink, lack of sleep other activities or things participants feel are related to the onset of arrhythmias
Association of available blood tests results to predict the risk of atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 3 months prior to 3 months after inclusion
  Blood tests may be useful in determining the effect of concomitant illness, their exacerbations, or, conversely, the stable course of the disease on the arrhythmia.
  Available results of each separate test (potassium, sodium, magnesium, BNP, creatinine, glomerular filtration rate, lipid profile, c-reactive protein) in relation to atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a period of 3 months prior to 3 months after inclusion.
Association of sleep analysis data with atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 7 days
  Each participant will be given a sleeping mat to put under the mattress and data collected from it in relation to atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a monitoring period of 7 days.
  Measured separately as:
  Sleep Quality Index, Apnea Episodes, Snoring Episodes, Snoring (%), Sleep Duration (Hours), Regular Sleep, Sleep Depth, Sleep Breaks
Temporal relation between changes in blood pressure and atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 7 days
  The results from the 48-hour blood pressure measurements (ambulatory BPM Mobil-o-graph's data) and additional 5 days measurements (Withings BPM) will be used to describe temporal relation between changes in blood pressure and atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a monitoring period of 7 days. The temporal relation will be measured as a time of blood pressure rise/fall before arrhythmia occurrence personalized for each individual and generalized for groups of individuals.
  Collected data:
  date, time, systole mean arterial pressure, Diastole, Peripheral pulse pressure (pPP), Heart rate (Hr), cSPB, cDBP, MAP-C2 (calibration for calculating the aortic central systolic blood pressure)
Association of echocardiographic results to predict the risk of atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 3 months prior to 3 months after inclusion.
  Echocardiography parameters will show cardiac status and function: chambers sizes, presence of left ventricular (LV) hypertrophy, atrial enlargement; the strains of left atrium and the predicted risk of these parameters in relation to atrial arrhythmias. Echocardiography will be acquired within a period of 3 months prior to 3 months after inclusion.
  Echocardiography parameters: Main: LV ejection fraction (LV EF) (%), LV end diastolic diameter (LVdd) (cm), Interventricular septal diameter (IVd) (cm), LV posterior wall diameter (LVPWd) (cm), E and A waves (m/s), Left atrial diameter (cm), LA volume index (ml/m2), LA maximum volume (ml), E' lat, E' med (cm/s), E' vid, E/e' vid, E deceleration time (ms). Additional parameters (%): mean contractile strain, 4 chamber (4 CH) contractile strain, 2 CH contractile strain, mean conduit strain, 4 CH conduit strain, 2 CH conduit strain, mean reservoir strain (%), 4 CH reservoir strain (%), 2 CH reservoir strain (%).
Association of parasympathetic and sympathetic tone to predict the risk of atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 7 days
  The activity of autonomic nervous system will be measured as heart rate variability (HRV), standard deviation of normal-to-normal heart rate intervals (SDNN) and other parameters in relation to atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a monitoring period of 7 days.
Association of physical activity to predict the risk of atrial arrhythmias in patients with previously diagnosed atrial fibrillation | 7 days
  To assess level of physical activity (measured as MET and the number of steps taken per day) in relation to atrial arrhythmias (atrial fibrillation, atrial flutter, atrial tachycardia, premature atrial contractions) within a monitoring period of 7 days.
Potential triggers named by participants, symptoms, burden of arrhythmia and the quality of life in patients with previously diagnosed atrial fibrillation before monitoring | 1 day
  Before the start of monitoring participants will fill out the questionnaire of most frequent known triggers, which could provoke their arrhythmias as well as mark the arrhythmia-related symptoms and the burden of arrhythmia in everyday life.
Usability of devices in everyday use | 1 day
  After the monitoring of 7 days participants will fill out the questionnaire of the convenience of each device and the willingness to use them if recommended by a physician in everyday practice.
Potential triggers named by participants, symptoms, burden of arrhythmia and the quality of life in patients with previously diagnosed atrial fibrillation after the collected information is presented to the patients | 3 months after the collected information is presented to the patient
  At least 3 months after the collected monitoring results are presented to the patients, the participants will fill out the questionnaire about changes of perceived potential triggers, symptoms, burden of arrhythmia and the quality of life ad symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Santaros Clinics, Vilnius, Vilniaus, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided